CLINICAL TRIAL: NCT01389713
Title: Patients With Reduced Ovarian Reserve and In Vitro Fertilization (IVF) Cycles. A Randomized Multicentric Comparison of a Protocol With High Doses of Gonadotropins and a Protocol With Clomiphene Citrate Only. Evaluation of Clinical Effectiveness and Economic Issues
Brief Title: Clomifene Citrate as First Line Treatment in in Vitro Fertilization Cycles for Patients With Lower Ovarian Reserve
Acronym: clomid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Istituto Clinico Humanitas (Other); IRCCS San Raffaele (Other); Istituti Clinici Zucchi (Other)
Responsible Party: Guido Ragni, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: clomid re-007
Record Dates: First submitted 2011-07-01; First posted 2011-07-08 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Infertility
Keywords: ovarian reserve; ovarian stimulation; clomifene citrate; high doses Follicle Stimulating Hormone (FSH)
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Gonadotropin-Releasing Hormone; Triptorelin Pamoate; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High doses (Active Comparator): Administration of high doses of gonadotrophins to stimulate ovarian follicular growth
  Interventions: Drug: GnRH analog and recombinant human FSH
- Clomid (Experimental): Administration of Clomiphene Citrate to obtain ovarian follicular growth
  Interventions: Drug: Clomifene Citrate

INTERVENTIONS:
Drug: Clomifene Citrate — 3x50 mg die for 5 days from day 3 to day 7 of the menstrual cycle
  Other Names: clomid
  Arms: Clomid
Drug: GnRH analog and recombinant human FSH — daily subcutaneous 0.1 mg decapeptyl from day 1-2 of the menstrual cycle and recombinant human FSH 450 IU/die from day 3.
  Other Names: decapeptyl; Gonal-F
  Arms: High doses

SUMMARY:
Women with compromised ovarian reserve requiring in vitro fertilization (IVF) still represent a demanding challenge for clinicians. It has classically been claimed that using higher dosages of gonadotropins may overcome the scarce ovarian responsiveness to hyper-simulation and increase the chances of success. However, scientific evidence supporting this view is scanty and costs are inevitably much higher. In this study, the investigators hypothesized that similar chances of pregnancy may be achieved with a mild stimulation using exclusively Clomiphene citrate (CC).

ELIGIBILITY:
Inclusion Criteria:

* age 18-42 years
* infertility status
* Day 3 serum FSH > 12 IU/ml in at least two occasions or previous poor response (≤3 oocytes retrieved) to hyper-stimulation

Exclusion Criteria:

* contraindications to infertility treatments or pregnancy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 289 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
live birth rate | end of the study (28 months)
  general "Live birth rate" will be recorded at the end of the study when all participants have performed their In vitro Fertilization (IVF) treatment.
  Live birth rate per single patients will be recorded 4 weeks after embryo transfer when a intrauterine gestational sac is expected to be seen in case of pregnancy.

SECONDARY OUTCOMES:
ratio pregnancies/costs | end of the study (28 months)
  at the end of the study the number of obtained pregnancies will be divided by the total costs of treatments in two groups. A cost in euros will be therefore estimated for every single pregnancy in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: guido ragni, md, Principal Investigator — Fondazione Ca' Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] Heijnen EM, Eijkemans MJ, De Klerk C, Polinder S, Beckers NG, Klinkert ER, Broekmans FJ, Passchier J, Te Velde ER, Macklon NS, Fauser BC. A mild treatment strategy for in-vitro fertilisation: a randomised non-inferiority trial. Lancet. 2007 Mar 3;369(9563):743-749. doi: 10.1016/S0140-6736(07)60360-2. PMID 17336650
- [Background] Eijkemans MJ, Heijnen EM, de Klerk C, Habbema JD, Fauser BC. Comparison of different treatment strategies in IVF with cumulative live birth over a given period of time as the primary end-point: methodological considerations on a randomized controlled non-inferiority trial. Hum Reprod. 2006 Feb;21(2):344-51. doi: 10.1093/humrep/dei332. Epub 2005 Oct 20. PMID 16239317
- [Derived] Ragni G, Levi-Setti PE, Fadini R, Brigante C, Scarduelli C, Alagna F, Arfuso V, Mignini-Renzini M, Candiani M, Paffoni A, Somigliana E. Clomiphene citrate versus high doses of gonadotropins for in vitro fertilisation in women with compromised ovarian reserve: a randomised controlled non-inferiority trial. Reprod Biol Endocrinol. 2012 Dec 18;10:114. doi: 10.1186/1477-7827-10-114. PMID 23249758